CLINICAL TRIAL: NCT01020734
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Acute Myelogenous Leukemia in Remission Using HLA-Matched Sibling Donors, HLA-Matched Unrelated Donors, or HLA-Mismatched Familial Donors - A Phase 2 Study
Brief Title: Donor Stem Cell Transplant or Bone Marrow Transplant in Treating Patients With Acute Myeloid Leukemia in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor of Internal Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000659891; AMC-UUCM-2009-0579
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with t(16;16)(p13;q22); recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); childhood acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute erythroleukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transplantation (Experimental): perform allogeneic HCT for patients with AML in CR1; then analyze various pre-transplantation variable, including donor type, for correlation to outcomes
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: methotrexate
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and methotrexate before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor stem cell transplant or bone marrow transplant works in treating patients with acute myeloid leukemia in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of allogeneic hematopoietic stem cell transplantation (HSCT) or bone marrow transplantation (BMT) from a HLA-matched sibling donor, HLA-matched unrelated donor, or HLA-mismatched familial donor, in terms of the frequency of relapse and duration of remission, in patients with acute myeloid leukemia (AML) who have either achieved complete remission (CR1) after induction chemotherapy or who experienced recurrent AML then achieved second CR (CR2) after salvage chemotherapy.

Secondary

* Determine the engraftment, donor chimerism, and secondary graft failure in these patients.
* Assess acute and chronic graft-vs-host disease, immune recovery, and infections in these patients.
* Determine transplantation-related mortality, leukemia-free survival, and overall survival of these patients.

OUTLINE:

* Conditioning chemotherapy and allogeneic bone marrow or hematopoietic stem cell transplantation (HSCT): After completion of induction chemotherapy and a resulting complete response (CR1) or salvage chemotherapy resulting in CR2, patients receive 1 of the following conditioning regimens and transplantations determined by age, co-morbidity, and type of available donor:

  * 15 to 55 years of age without significant co-morbidity* undergoing HLA-matched sibling bone marrow transplantation (BMT) (BuCy conditioning): Patients receive busulfan IV once daily on days -7 to -4 and cyclophosphamide IV over 1-2 hours once daily on days -3 and -2. Patients then undergo an allogeneic BMT on day 0.
  * Older than 55 years or younger than 55 years with co-morbidity* undergoing HLA-matched sibling BMT; patients of any age undergoing HLA-matched unrelated HSCT; and for patients of any age undergoing HLA-mismatched familial donor HSCT (BuFluATG conditioning): Patients receive busulfan IV once daily on days -7 and -6, fludarabine phosphate IV over 30 minutes once daily on days -7 to -2, anti-thymocyte globulin IV over 4 hours once daily on days -3 to -1, and methylprednisolone IV over 30 minutes once daily on days -4 to -1. Patients then undergo either an allogeneic BMT on day 0 or allogeneic peripheral blood hematopoietic stem cell infusions on days 0-1 or 0-2.

NOTE: *Significant co-morbidity is defined as residual fungal or other infections in the lung or other viscera and residual organ toxicities occurring during induction or consolidation chemotherapy.

* GVHD prophylaxis: Patients receive cyclosporine orally or IV over 2-4 hours twice daily beginning on day -1 followed by a taper starting on day 30 (BuFluATG conditioning) or day 60 (BuCy conditioning). Patients also receive methotrexate IV on days 1, 3, and 6 after the last day of donor cell infusion.
* CNS prophylaxis: Patients receive intrathecal (IT) methotrexate once before conditioning regimen. Patients receive IT methotrexate once every 2 weeks for 3 times after transplantation and platelet recovery. Patients also receive leucovorin calcium orally or IV over 4 hours after IT methotrexate and then once every 6 hours for a total of 8 doses after each dose of IT methotrexate.

After completion of study therapy, patients are followed every 3 months for 3 years and then annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) meeting 1 of the following criteria:

  * Achieved complete response (CR1) after induction chemotherapy
  * Recurrent AML that went into second CR (CR2) after salvage chemotherapy, except those who have undergone prior allogeneic HSCT
* No acute promyelocytic leukemia or acute myeloid leukemia with chromosomal changes t(8;21), inv 16, or t(15;17)
* Must have a donor available meeting one of the following criteria:

  * HLA-matched sibling of 65 years or younger
  * 6/6 HLA-matched unrelated donor (younger than 55 years) for antigen A, B, and DR
  * HLA-mismatched family member (offspring, parents, haploidentical sibling)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 2.0 mg/dL
* AST < 3 times the upper limit of normal
* Creatinine < 2.0 mg/dL
* Ejection fraction > 40% on MUGA scan
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2011-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of the treatment measured in terms of frequency of relapse and duration of remission | up to 2 years after transplantation
  duration of CR, leukemia recurrence

SECONDARY OUTCOMES:
Engraftment | up to 35 days after transplantation
  achievement of neutrophil count over 500/ul
Acute and chronic graft-versus-host disease | up to 100 days for acute GVHD and up to 2 years for chronic GVHD
Treatment-related mortality | up to 2 years after transplantation
Leukemia-free survival and overall survival | up to 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Inje University - Haeundae Paik Hospital, Busan
  - Asan Medical Center - University of Ulsan College of Medicine, Seoul